CLINICAL TRIAL: NCT03645863
Title: A Clinical Pharmacological Study to Evaluate the Effects of Iron Supplements on the Pharmacokinetics of MT-6548 in Healthy Male Volunteers
Brief Title: Effects of Iron Supplements on the Pharmacokinetics of MT-6548
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MT-6548-J05
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Healthy
MeSH Terms: interventions — vadadustat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1 (Experimental): Subject will receive MT-6548 on Day 1, 4, and 7. Subject will receive Iron supplement A on Day 1, 4, or 7. Subject will receive Iron supplement B on Day 1, 4, or 7.
  Interventions: Drug: MT-6548; Drug: Iron supplement A; Drug: Iron supplement B
- Cohort 2 (Experimental): Subject will receive MT-6548 on Day 1 and 4. Subject will receive Iron supplement C on Day 1 or 4.
  Interventions: Drug: MT-6548; Drug: Iron supplement C
- Cohort 3 (Experimental): Subject will receive MT-6548 on Day 1 and 4. Subject will receive Iron supplement D on Day 1 or 4.
  Interventions: Drug: MT-6548; Drug: Iron supplement D

INTERVENTIONS:
Drug: MT-6548 — Oral tablet
  Other Names: vadadustat; AKB-6548
Drug: Iron supplement A — Oral tablet
  Arms: Cohort 1
Drug: Iron supplement B — Oral tablet
  Arms: Cohort 1
Drug: Iron supplement C — Oral tablet
  Arms: Cohort 2
Drug: Iron supplement D — Oral tablet
  Arms: Cohort 3

SUMMARY:
The objectives of this study are to investigate the pharmacokinetics and safety of MT-6548 co-administered with iron supplements in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Parents and each grandparent of subjects are Japanese
* Subjects judged as appropriate for this study by investigators based on the results of the tests at Screening, Day -1 and Day 1

Exclusion Criteria:

* Subjects with signs of heart diseases on the result of screening test
* Subjects with current conditions or histories of drug addiction or alcohol addiction
* Subjects judged by investigators that they cannot comply with the prohibition during the confinement period
* Subjects who have taken MT-6548 before
* Subjects with current conditions or histories of drug or food allergies
* Subjects with BMI below18.5 kg/m2, BMI above 25.0 kg/m2 or body weight below 50.0 kg at the screening test
* Subjects who have undergone platelet or plasma donation 2 weeks prior to the consent
* Subjects who have undergone blood donation or blood draw of 400 mL or above within 12 weeks prior to the consent, or 200 mL or above within 4 weeks prior to the consent
* Subjects who have undergone blood donation or blood draw of 800 mL or above within one year prior to the consent
* Subjects who have undergone surgical operations that can affect gastrointestinal absorption of medication (appendectomy and hernioplasty do not meet this exclusion criterion)
* Subjects with positive results for HBs antigen, syphilis serum reaction, HCV antibody or HIV antigen / antibody at the screening test
* Subjects who are unwilling to consent to use contraception from the beginning of study period to 90 days following the final dose of the study drug
* Subjects who have participated in another clinical study and received study drugs within 12 weeks prior to consent, or within 5 times the half-life of the study drug (whichever is longer)
* Subjects who have taken any medications except for the drug used for this clinical study within 7 days prior to the first dose of the study drug
* Subjects who have had supplements within 7 days prior to the first dose of the study drug
* Subjects who have had apples, citrus fruits such as grapefruits or any food products that contain apples or citrus fruits within 7 days prior to the first dose of the study drug
* Subjects who have had food products which contain St John's Wort within 2 weeks prior to the first dose of the study drug

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Research site, Tokyo, Japan

REFERENCES:
- [Result] Kokado Y, Kawai K, Nanjo T, Kinoshita S, Kondo K. In Vitro and Clinical Pharmacokinetic Studies of the Effects of Iron-containing Agents on Vadadustat, an Oral Hypoxia-inducible Factor-Prolyl Hydroxylase Inhibitor. Clin Ther. 2021 Aug;43(8):1408-1418.e5. doi: 10.1016/j.clinthera.2021.06.013. Epub 2021 Sep 10. PMID 34511184

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Subject will receive oral MT-6548 tablet (150 mg) on Day 1, 4, and 7. Subject will receive Iron supplement A (Ferric Citrate Hydrate 250 mg) on Day 1, 4, or 7. Subject will receive Iron supplement B (Sodium Ferrous Citrate 50 mg) on Day 1, 4, or 7.
- Cohort 2: Subject will receive oral MT-6548 tablet (150 mg) on Day 1 and 4. Subject will receive Iron supplement C (Sucroferric oxyhydroxide 500 mg) on Day 1 or 4.
- Cohort 3: Subject will receive MT-6548 on Day 1 and 4. Subject will receive Iron supplement D (Dried Ferrous Sulfate 105 mg) on Day 1 or 4.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 21 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 21 | 20 | 20 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 20 | 61
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 21 | 20 | 20 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 21 | 20 | 20 | 61
  Other | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity(AUC0-∞) of Unchanged MT-6548
Time Frame: Up to Day 8 (Cohort 1), Up to Day 5 (Cohort 2, 3)
Population: This analysis was performed only in subjects who have the data at each visit.
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 21 | 20 | 20
ug*h/mL
  MT-6548 | 105.3 (17.0) | 100.2 (12.4) | 129.3 (18.1)
  MT-6548+Iron supplement A: number analyzed (Participants) | 20 | 0 | 0
  MT-6548+Iron supplement A | 49.2 (16.9) |  |
  MT-6548+Iron supplement B: number analyzed (Participants) | 20 | 0 | 0
  MT-6548+Iron supplement B | 37.2 (19.5) |  |
  MT-6548+Iron supplement C: number analyzed (Participants) | 0 | 20 | 0
  MT-6548+Iron supplement C |  | 47.7 (13.9) |
  MT-6548+Iron supplement D: number analyzed (Participants) | 0 | 0 | 20
  MT-6548+Iron supplement D |  |  | 16.0 (10.7)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Unchanged MT-6548
Time Frame: Up to Day 8 (Cohort 1), Up to Day 5 (Cohort 2, 3)
Population: This analysis was performed only in subjects who have the data at each visit.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 21 | 20 | 20
ug/mL
  MT-6548 | 14.5 (2.61) | 15.5 (2.83) | 27.1 (5.93)
  MT-6548+Iron supplement A: number analyzed (Participants) | 20 | 0 | 0
  MT-6548+Iron supplement A | 7.76 (3.93) |  |
  MT-6548+Iron supplement B: number analyzed (Participants) | 20 | 0 | 0
  MT-6548+Iron supplement B | 5.96 (3.09) |  |
  MT-6548+Iron supplement C: number analyzed (Participants) | 0 | 20 | 0
  MT-6548+Iron supplement C |  | 9.37 (3.21) |
  MT-6548+Iron supplement D: number analyzed (Participants) | 0 | 0 | 20
  MT-6548+Iron supplement D |  |  | 2.65 (1.95)

3. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Unchanged MT-6548
Time Frame: Up to Day 8 (Cohort 1), Up to Day 5 (Cohort 2, 3)
Population: This analysis was performed only in subjects who have the data at each visit.
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 21 | 20 | 20
h
  MT-6548 | 3.00 [1.50 to 5.00] | 1.00 [0.50 to 5.00] | 2.00 [1.00 to 3.00]
  MT-6548+Iron supplement A: number analyzed (Participants) | 20 | 0 | 0
  MT-6548+Iron supplement A | 3.00 [1.00 to 6.00] |  |
  MT-6548+Iron supplement B: number analyzed (Participants) | 20 | 0 | 0
  MT-6548+Iron supplement B | 4.00 [1.00 to 5.00] |  |
  MT-6548+Iron supplement C: number analyzed (Participants) | 0 | 20 | 0
  MT-6548+Iron supplement C |  | 1.00 [0.50 to 3.00] |
  MT-6548+Iron supplement D: number analyzed (Participants) | 0 | 0 | 20
  MT-6548+Iron supplement D |  |  | 3.00 [0.50 to 5.00]

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Until the Last Quantifiable Concentration (AUC0-last) of Unchanged MT-6548
Time Frame: Up to Day 8 (Cohort 1), Up to Day 5 (Cohort 2, 3)
Population: This analysis was performed only in subjects who have the data at each visit.
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 21 | 20 | 20
ug*h/mL
  MT-6548 | 100.4 (16.1) | 96.3 (11.7) | 125 (17.2)
  MT-6548+Iron supplement A: number analyzed (Participants) | 20 | 0 | 0
  MT-6548+Iron supplement A | 47 (16.6) |  |
  MT-6548+Iron supplement B: number analyzed (Participants) | 20 | 0 | 0
  MT-6548+Iron supplement B | 36 (19.1) |  |
  MT-6548+Iron supplement C: number analyzed (Participants) | 0 | 20 | 0
  MT-6548+Iron supplement C |  | 46.4 (13.6) |
  MT-6548+Iron supplement D: number analyzed (Participants) | 0 | 0 | 20
  MT-6548+Iron supplement D |  |  | 14.9 (10.4)

5. Primary Outcome: Mean Residence Time From Zero to Infinity (MRT0-∞) of Unchanged MT-6548
Time Frame: Up to Day 8 (Cohort 1), Up to Day 5 (Cohort 2, 3)
Population: This analysis was performed only in subjects who have the data at each visit.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 21 | 20 | 20
h
  MT-6548 | 8.23 (0.95) | 6.97 (0.82) | 6.56 (1.05)
  MT-6548+Iron supplement A: number analyzed (Participants) | 20 | 0 | 0
  MT-6548+Iron supplement A | 8.06 (1.05) |  |
  MT-6548+Iron supplement B: number analyzed (Participants) | 20 | 0 | 0
  MT-6548+Iron supplement B | 7.28 (0.98) |  |
  MT-6548+Iron supplement C: number analyzed (Participants) | 0 | 20 | 0
  MT-6548+Iron supplement C |  | 5.76 (0.86) |
  MT-6548+Iron supplement D: number analyzed (Participants) | 0 | 0 | 20
  MT-6548+Iron supplement D |  |  | 7.21 (1.47)

6. Primary Outcome: Apparent Terminal Elimination Rate Constant (Kel) of Unchanged MT-6548
Time Frame: Up to Day 8 (Cohort 1), Up to Day 5 (Cohort 2, 3)
Population: This analysis was performed only in subjects who have the data at each visit.
Measure: Mean (Standard Deviation); unit: /h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 21 | 20 | 20
/h
  MT-6548 | 0.1314 (0.0181) | 0.1356 (0.0216) | 0.1354 (0.0194)
  MT-6548+Iron supplement A: number analyzed (Participants) | 20 | 0 | 0
  MT-6548+Iron supplement A | 0.1302 (0.0146) |  |
  MT-6548+Iron supplement B: number analyzed (Participants) | 20 | 0 | 0
  MT-6548+Iron supplement B | 0.1647 (0.0295) |  |
  MT-6548+Iron supplement C: number analyzed (Participants) | 0 | 20 | 0
  MT-6548+Iron supplement C |  | 0.1629 (0.031) |
  MT-6548+Iron supplement D: number analyzed (Participants) | 0 | 0 | 20
  MT-6548+Iron supplement D |  |  | 0.1518 (0.0499)

7. Primary Outcome: Terminal Elimination Half-life (t1/2) of Unchanged MT-6548
Time Frame: Up to Day 8 (Cohort 1), Up to Day 5 (Cohort 2, 3)
Population: This analysis was performed only in subjects who have the data at each visit.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 21 | 20 | 20
h
  MT-6548 | 5.38 (0.8) | 5.22 (0.75) | 5.23 (0.83)
  MT-6548+Iron supplement A: number analyzed (Participants) | 20 | 0 | 0
  MT-6548+Iron supplement A | 5.39 (0.61) |  |
  MT-6548+Iron supplement B: number analyzed (Participants) | 20 | 0 | 0
  MT-6548+Iron supplement B | 4.33 (0.71) |  |
  MT-6548+Iron supplement C: number analyzed (Participants) | 0 | 20 | 0
  MT-6548+Iron supplement C |  | 4.4 (0.86) |
  MT-6548+Iron supplement D: number analyzed (Participants) | 0 | 0 | 20
  MT-6548+Iron supplement D |  |  | 5.05 (1.63)

ADVERSE EVENTS:
Time Frame: Day 1 to 10 (cohort 1), Day 1 to 7 (cohort 2 and 3)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 4/21 | 0/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=21) | Cohort 2 (N=20) | Cohort 3 (N=20)
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT03645863/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT03645863/SAP_001.pdf